CLINICAL TRIAL: NCT03412903
Title: The Pharmacist in the Acute Geriatric Inpatient Treatment Team - Impact on Re-hospitalization and Trans-sectoral Communication
Brief Title: The Pharmacist in the Acute Geriatric Inpatient Treatment Team
Acronym: AGITATE
Status: Completed | Type: Observational
Sponsor: Prof. Dr. med. Cornelius Bollheimer (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Cornelius Bollheimer, Univ.-Prof. Dr. med., Klinikdirektor, RWTH Aachen University
Organization: RWTH Aachen University (Other)
Other Study IDs: 17-137; EK 230/17 (Other: Ethics Committee at the RWTH Aachen Faculty of Medicine)
Record Dates: First submitted 2018-01-19; First posted 2018-01-29 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Pharmacists in Geriatric Health Services; Conditions Unspecified
Keywords: Acute geriatric treatment; Inpatient treatment team; Elderly; Pharmacist; Comprehensive pharmaceutical assessment; Medication history; Medication reconciliation; Adherence; Medication therapy management; Pharmaceutical consultation; Drug-Related Side Effects and Adverse Reactions; Drug interactions; Pharmaceutical Council; Drug regime acceptance; Patient Care Team; Hospital Pharmacy Service; Polypharmacy; Hospitalization; Pharmaceutical Services
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: First observational period: Standard care without an advising pharmacist, 140 patients
- Implementation group: Second observational period: Standard care with an advising pharmacist, 140 patients
- Learning success group: Second observational period: Standard care without an advising pharmacist, 30 patients

SUMMARY:
This trial investigates the effects of a comprehensive pharmaceutical assessment in an acute care geriatric hospital on the number of hospital readmissions and patient's days spent at home.

DETAILED DESCRIPTION:
Drug-related problems are common in elderly patients. These problems can not only be regarded from a medical or economical point of view (i.e. hospitalization, drug related deaths, longer hospital stays and increased healthcare costs) but also from a patient centered perspective: Drug therapy may not be sufficiently explained by health care practitioners, patients might suffer from side effects, the number of different medications could be too large and their intake schedule too difficult, all of this leading to a reduced adherence. In addition, medication histories are rarely accurate in older patients and doctor's letters do not always meet the requirements of a complex drug therapy. At the transition from inpatient to outpatient treatment this can lead to a significant loss of information and subsequently cause patient harm.

In Germany, clinical, ward-based pharmacists are not yet established in contrast to other countries (i.e. Great Britain, Canada and Australia). However, the implementation of a clinical pharmacist may particularly address the problems described above. The present study therefore describes the implementation of a comprehensive pharmaceutical assessment in an acute care geriatric hospital.

The above mentioned pharmaceutical assessment consists of the following steps:

First, the pharmacist will obtain the patient's medication history following the protocol of "best possible medication history" (WHO). Furthermore, he will ascertain the patient's adherence to his/her drug regime. With the information obtained, he will then carry out a thorough medication review (regarding interactions, contraindications, suitability for the elderly, dosage regimes, etc.) in order to develop a suggestion for the best possible drug regime, which is discussed with the treating physician. In addition, he will also observe possible side effects and provide information on the background and significance of every single drug to the patient and/or his/her care-giver. Furthermore, the handling of difficult devices (i.e. insulin pens, inhalators and transdermal therapeutic systems) will be individually explained. Finally, the pharmacist will prepare a distinctive paragraph in the medical discharge report in which he explains the changes in the medication regime during the inpatient period to the general practitioner and will also elaborate possible interactions and problems concerning the patient's medication (pharmaceutical council).

The main outcome to be evaluated will be the number of hospital readmissions and drug related hospital readmissions within six months after discharge (recorded at one, three and six months). The secondary outcome will be the days spent at home (also recorded at one, three and six months), time to readmission, changes in medication within six months and the acceptance of the supposed medication regime by the general practitioner (GP).

The study will be conducted as a before and after comparison in which the steps described above will be implemented successively: In the first phase (140 patients planned for an observation period of eight months), patients will receive standard care and the pharmacist will only obtain the medication history shortly after admission. Results and discrepancies will be discussed with the attending physician of the hospital. After discharge, described outcomes will be documented. In the second phase (140 patients planned for an observation period of eight months), the pharmacist will conduct all of the activities described above. The outcomes will be documented as in phase one.

We expect that the comprehensive pharmaceutical assessment in the second phase will lead to a better coordination regarding the medication regime, enhance the patient's knowledge of their medication, thus improving their adherence to the therapy and that the pharmaceutical council will ensure a better trans-sectoral communication to the GP with a higher acceptance of the supposed drug regime in the doctor's letter. All these improvements combined might reduce hospital readmissions and increase the patient's days spent at home.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric complex treatment (Operation and procedure code (German: "Operationen- und Prozedurenschlüssel", OPS) 8-550)
* In-patient stay for at least 7 days
* Written informed consent of the patient or the legal representative
* Existing concomitant drug therapy at the time of the inpatient admission

Exclusion Criteria:

* Patients, that were already included in the study beforehand
* Patients classified as terminally ill by the medical staff
* Patients, that are incapable to give their informed consent and who do not have a legal representative

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to the clinic for internal medicine and geriatrics of the Franziskus Hospital Aachen (chair of geriatrics and geriatric medicine of the RWTH Aachen University)
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Drug related re-hospitalization | 6 months
  Number of re-hospitalizations with causal relation to one or more medicinal products, to examine the potential effect of an advising pharmacist

SECONDARY OUTCOMES:
Overall re-hospitalization | 6 months
  Overall number of re-hospitalizations within the observational period per patient
Days spent at home | 6 months
  Number of days within the observational period not spent in a hospital, short-term care facility, rehabilitation centre, day-care hospital, emergency department or other medical facilities
Period of time until the potential re-hospitalization into the inpatient sector | 6 months
  Time between the discharge and a potential re-hospitalization per patient
Acceptance of the recommended medication plan by the further treating primary care physicians | 6 months
  Adoption of the medication plan, recommended in the doctor's letter, by the further treating primary care physicians
Time required for the pharmacists support | 6 months
  Expenditure of time, required for the pharmacists support, per patient within the implementation group
Completeness of the pharmaceutical anamnesis in the course of the inpatient admission | 6 months
  Comparison between the pharmaceutical anamnesis conducted by the doctor and the pharmacist, respectively
Evaluation of the clinical relevance of the medicinal products, which were not assessed by the doctors | 6 months
  The evaluation will be conducted by an interdisciplinary group using the focus group method.

CONTACTS AND LOCATIONS:
Overall Officials: Cornelius Bollheimer, Prof. Dr., Study Director — University Hospital, Aachen
Locations (1):
- Franziskushospital, Aachen, Northrheinwestfalia, Germany

IPD SHARING:
Plan to Share IPD: No